CLINICAL TRIAL: NCT07307937
Title: Movement Sonification as an add-on to Immediate Post-event Psychotherapeutic Intervention in the Management of Acute Stress Disorder: a Feasibility and Acceptability Study
Acronym: SONICUMP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: APHP241593
Record Dates: First submitted 2025-08-20; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-09

CONDITIONS: Acute Stress Disorder Symptoms
Keywords: post-traumatic stress disorder; potentially traumatic events; transforming the patient's movement into sound information
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sonification (Experimental): The sonification of movement is an act studied in this research.
  Interventions: Device: The sonification of movement is an act studied in this research.

INTERVENTIONS:
Device: The sonification of movement is an act studied in this research. — The sonification of movement is an act studied in this research at visit 1, visit 2 and visit 3

SUMMARY:
Natural disasters, conflicts, persecution, population displacement, often traumatic migration experiences, and terrorist attacks are all factors that currently expose a significant proportion of the world's population to potentially traumatic events (PTEs). When a person is exposed to a PTE, symptoms of acute stress disorder (ASD) may occur in the immediate aftermath of the PTB, i.e., within the month following the event. These symptoms are dominated by dissociation, which includes depersonalization, i.e., the feeling of being disconnected from one's body. Managing these symptoms can prevent the subsequent onset of post-traumatic stress disorder (PTSD), a serious illness and public health concern. The recommended treatment combines an immediate post-event psychotherapeutic intervention (IPPI) and, where appropriate, medication with anxiolytics from the antihistamine class or antipsychotics

DETAILED DESCRIPTION:
In France, IPPI is carried out by the medical-psychological emergency units (CUMP) in each department. Patients are referred to these units by the CUMPs themselves when they are called out by the SAMU (emergency medical service) to the scene of mass accidents (attacks, fires, suicides in public places, etc.), or by departmental doctors and medico-legal emergency services for individual EPTs (sexual or physical assault, etc.). In Seine-Saint-Denis, the CUMP 93 receives 60 to 100 patients per year in the immediate post-traumatic phase.

The purpose of IPPI is to reconnect the traumatic experience with known representations. These interventions have demonstrated effectiveness,although their preventive impact on PTSD remains limited. Movement sonification is an augmented auditory reality technique that transforms a patient's movements into sound through connected wristbands and a speaker system. By enriching bodily perception, this technique may enhance the efficacy of trauma-focused psychotherapies.

This study aims to assess the acceptability and feasibility of using movement sonification in combination with IPPI for the treatment of ASD. It thereby addresses an urgent need for primary prevention of PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over
* Who have experienced a potentially traumatic event (PTE) other than the death of a loved one
* Who have been referred to the medical-psychological emergency unit (CUMP 93) within one month of the PTE
* Who are experiencing acute stress disorder (ASD) according to DSM-5 criteria
* Have health insurance
* Have signed a written informed consent form

Exclusion Criteria:

* Severe motor impairment rendering the use of sonification technology impractical
* Deaf, mute, or hearing-impaired patients
* Adults under guardianship or conservatorship, under judicial protection, or deprived of liberty
* Suffering from chronic psychotic disorder or bipolar disorder
* Central neurological disease defined by a medical report (including brain damage, cortical or subcortical atrophy, dementia, stroke, transient ischemic attack, head trauma, epilepsy, or seizure)
* Presenting a proven severe risk of suicide
* Substance use disorder (excluding tobacco)
* Pregnant or breastfeeding women
* Participation in another interventional study on ESA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the feasibility of movement sonification in association with IPPI in the treatment of ESA. | 6 weeks
  Success rate, defined as an individual adherence rate of at least two sessions completed with movement sonification out of the three sessions planned.

SECONDARY OUTCOMES:
Dissociative symptoms | 6 weeks
  1) Change in the severity of dissociative symptoms assessed by:
  1a) • Clinician-Administered Dissociative States Scale from V1 to V4. A high score on the Clinician-Administered Dissociative States Scale (range 0 to 92) indicates a more severe degree of dissociative symptoms.
Dissociative symptoms | 6 weeks
  1) Change in the severity of dissociative symptoms assessed by:
  1b)• Multidimensional Assessment of Interoceptive Awareness-2 at V1 and V4. A high score on the Multidimensional Assessment of Interoceptive Awareness-2 (range 0 to 160) reflects more developed interoceptive awareness, with an increased ability to recognize and respond adaptively to bodily sensations.
Agency (sense of control over the external environment) | 6 weeks
  Changes in agency assessed by the Fribourg Sense of Agency Scale from V1 to V4. A high score on the Fribourg Sense of Agency Scale (range 13 to 91) is associated with an increased perception of personal control and a stronger integration of conscious action with personal responsibility.
The overall clinical response | 6 weeks
  Change in clinical impression assessed by the Clinical Global Impression-Severity from V1 to V4. The scale ranges from 1 to 7, where a low value indicates no symptoms and 7 indicates a terminal stage disorder.
The overall clinical response | 6 weeks
  Change in clinical impression assessed by Clinical Global Impression-Improvement from V2 to V4. The scale ranges from 1 to 7, where a low value represents significant improvement and 7 indicates considerable deterioration.
Overall functioning | 6 weeks
  Change in overall functioning assessed by the Global Assessment of Functioning from Visit 1 to Visit 4.
  The Global Assessment of Functioning, scale is used to rate how serious a mental illness may be. It measures how much a person's symptoms affect their day-to-day life on a scale of 0 to 100.A high score on the Global Assessment of Functioning suggests very good or near-normal overall functioning.
Symptoms associated with ESA in patients with initial symptoms of traumatic dissociation, compared to those without | 6 weeks
  Comparison of changes in scale between patients according to the level of dissociation assessed by the Clinician-Administered Dissociative States Scale. A high score on the Clinician-Administered Dissociative States Scale (range 0 to 92) indicates a more severe degree of dissociative symptoms.
Symptoms associated with ESA in patients with initial symptoms of traumatic dissociation, compared to those without | 6 weeks
  Comparison of changes in scale between patients according to the level of dissociation assessed by the Multidimensional Assessment of Interoceptive Awareness 2. A high score on the Multidimensional Assessment of Interoceptive Awareness 2 (range 0 to 160) reflects more developed interoceptive awareness, with an increased ability to recognize and respond adaptively to bodily sensations.
Symptoms associated with ESA in patients with initial symptoms of traumatic dissociation, compared to those without | 6 weeks
  Comparison of changes in scale between patients according to the level of dissociation assessed by Fribourg Sense of Agency Scale. A high score on the Fribourg Sense of Agency Scale (range 13 to 91) is associated with an increased perception of personal control and a stronger integration of conscious action with personal responsibility.
Symptoms associated with ESA in patients with initial symptoms of traumatic dissociation, compared to those without | 6 weeks
  Comparison of changes in scale between patients according to the level of dissociation assessed by the Global Impression-Severity. The scale ranges from 1 to 7, where a low value indicates no symptoms, and 7 indicates a terminal condition.
Symptoms associated with ESA in patients with initial symptoms of traumatic dissociation, compared to those without | 6 weeks
  Comparison of changes in scale between patients according to the level of dissociation assessed by the Clinical Global Impression-Improvement. The scale ranges from 1 to 7, where a low value represents a significant improvement, and 7 indicates a considerable deterioration.
Symptoms associated with ESA in patients with initial symptoms of traumatic dissociation, compared to those without | 6 weeks
  Comparison of changes in scale between patients according to the level of dissociation assessed by the Global Assessment Functioning. A high Global Assessment of Functioning score (range from 0 to 100) suggests very good or near-normal overall functioning.
Evaluate the experience and acceptability of patients and caregivers (qualitative analysis). | 6 weeks
  The evaluation of the experience and acceptability will be carried out using a semi-structured interview with the patient at Visit 4

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Avicenne, Bobigny, France

IPD SHARING:
Plan to Share IPD: No